CLINICAL TRIAL: NCT05098886
Title: An Open Label, Randomized, Single Dose, Crossover Study to Evaluate the Pharmacokinetics and Safety of DA-5210 10/1000mg in Healthy Subjects at Fed State
Brief Title: Phamacokinetics and Safety Profiles of DA-5210 10/1000mg in Healthy Subjects at Fed State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIBE2021-54
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental)
  Interventions: Drug: DA-5210 10/1000mg; Drug: DA-5210-R 10/1000mg
- Sequence B (Experimental)
  Interventions: Drug: DA-5210 10/1000mg; Drug: DA-5210-R 10/1000mg

INTERVENTIONS:
Drug: DA-5210 10/1000mg — single dose administration (one tablet once a day)
Drug: DA-5210-R 10/1000mg — single dose administration (one tablet once a day)

SUMMARY:
Phamacokinetics and safety profiles of DA-5210 10/1000mg in Healthy subjects at Fed State

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* BMI between 18 and 30 kg/m2
* Body weight : Male≥50kg, Female≥45kg

Exclusion Criteria:

* Allergy or Drug hypersensitivity
* Clinically significant Medical History

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-07 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
AUCt | pre-dose~48 hours post-dose
  area under the curve
Cmax | pre-dose~48 hours post-dose
  maximum plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea